CLINICAL TRIAL: NCT00267995
Title: Proposal for Retrospective Review of Ross Aortic Valve Replacement Patients
Brief Title: Ross Aortic Valve Replacement Patients
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Kirk R Kanter, MD, Children's Healthcare of Atlanta
Other Study IDs: 03-047
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: Pediatric; cardiac; Ross procedure; Aortic valve replacement; Proximal buttressing technique
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Ross procedure has become the surgery of choice for aortic valve replacement in children. This consists of taking a child's own pulmonary valve (the autograft) and replacing the child's diseased aortic valve with the autograft. At times, this can involve either enlarging or reducing the diameter of the aortic annulus to make the valve fit properly. The patient's own pulmonary valve is then replaced, most typically with a human heart valve (a homograft). There has been some concern in the literature that as time goes on, the autograft will dilate and the patient will develop progressive aortic insufficiency.

Since 1994, we have performed almost 50 Ross procedures in children and young adults. Contrary to many reports from the literature, we have not recognized a problem with autograft enlargement and progressive aortic insufficiency. One thing that we have done differently from other centers is that we have modified the insertion technique of the autograft into the native aortic root. This involves a second buttressing suture layer. Not only does this have the immediate effect of reducing bleeding complications, we postulate that it has the long-term effect of stabilizing the autograft and preventing aortic root dilatation.

We hypothesize that this proximal buttressing technique for the Ross procedure has a two-fold benefit. Firstly, it reduces the amount of bleeding in the postoperative period. Secondly, it prevents late autograft root dilatation.

DETAILED DESCRIPTION:
This is a retrospective chart review examining our experience with the Ross procedure. There will be a treatment and control group. The treatment group will be children who have had the Ross procedure with the proximal buttressing technique. The control or comparisons group would be Ross procedure patients who did not receive the proximal buttressing technique. All children's charts reviewed will be of patients who had their surgery at Children's Healthcare of Atlanta between December 1994 and August 2003; only information available up until October 10, 2003 will be used for this study. We will review approximately 75 charts for this study.

The first aim of the study would be to examine basic information regarding bleeding incidence. The following information will be collected on both groups:

* Amount of chest tube bleeding within the first 24 hours, and
* Number of patients who required re-exploration for bleeding
* Time from cardiopulmonary bypass removal to time leaving the operating room (indicator of the need to "dry up").

The second aim of the study would be to review the echocardiograms on these patients. The pulmonary valve size before the Ross procedure would be measured on the preoperative transthoracic or transesophageal echocardiogram. This would then be compared with postoperative studies in the Operating Room by transesophageal echocardiography. The pre-discharge echocardiogram and follow-up echocardiograms (which are a routine for these patients and, therefore, would not be necessary to add to the study protocol) would be reviewed. Autograft root diameters would be measured. The diameters would be at the level of the valve leaflets, at the level of the commissures and at the sinotubular ridge. These would be compared against published Z values for these patients by age, weight and body surface area. At the same time, any degree of aortic insufficiency or left ventricular outflow tract obstruction would be noted and recorded. One non-invasive cardiologist will review all old echocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* Ross procedure with and without Proximal butressing technique
* Ross procedure between 12.1994 and 8.2003

Exclusion Criteria:

* those who do not meet inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Retro chart review
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 1994-12

CONTACTS AND LOCATIONS:
Overall Officials: Kirk R. Kanter, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States